CLINICAL TRIAL: NCT05624021
Title: Efficacy of Scapular Functional Training Combined With Isometric Exercises on Pain, Range of Motion, and Functions Among Individual With Mechanical Neck Pian
Brief Title: Effect of Functional Training and Isometric Exercises on Pain, ROM, and Functional Status in Patients With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Majmaah University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Prinicipal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2019-17
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Range of motion; Functional limitations; Isometric exercises; Functional training
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blinded study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFT group (Experimental): Received Scapular functional training and cervical isometric exercises
  Interventions: Other: Scapular functional training; Other: Cervical isometric exercises; Other: Moist heating
- Conventional group (Active Comparator): Received only isometric cervical exercises and heating
  Interventions: Other: Cervical isometric exercises; Other: Moist heating

INTERVENTIONS:
Other: Scapular functional training — The scapular functional training consists of press up and push up plus. Press up was done in sitting position on the training bench, feet on the floor with straight arm and the palms on the edge of the bench fingers pointing forward and then lift off and dip down just in front of the seat by moving the shoulder girdle. Progression is done by placing weight on the thigh. Push-up plus exercise started from a push up position on the hand, feet or knees and keeping the torso rigid by bracing the abdominals followed by protracting the scapula as high as possible. Progression is done moving from knees to the feet or adding resistance on the upper back. The training continued for three sessions per week for four weeks.
  Arms: SFT group
Other: Cervical isometric exercises — The isometric neck exercises taught to all the participants to perform in neutral sitting positions at home thrice a day for 15-days continuously. The sequences of exercises were shoulder circling in clockwise and anticlockwise direction, scapular retraction with cervical retraction, neck flexion, extension, either side of lateral bending/flexion, left and right rotation. Each exercise follows a set of 10 repetition of maximum voluntary contraction with a progressive hold time of 3, 5, 7, and 10 seconds depending on the severity of pain and tolerance of the participants.
Other: Moist heating — A hydrocollator moist heat packs was applied over back of the neck in supine position to receive optimal heating. It was given for 20 minutes/day, five-day a week for four-week.

SUMMARY:
Work-related musculoskeletal disorders have been rising fast around the globe leading to neck pain and scapular muscle dysfunction, contributing to a decrease in neck movements and functional limitations. This study aimed to determine the efficacy of scapular functional exercise (SFE) in combination with cervical isometric exercises (CIE) on neck pain, cervical range of motion, and functional limitations among participants with chronic mechanical neck pain.The study was based on a two-arm parallel group pretest-posttest randomized control trial design. Thirty participants (females 21 and males 9; average age 28.94±3.77 years) were randomly allocated to groups A and B (n=15/group). The group's A and B participants received a common intervention, such as CIE and hot packs. However, group A received the SFE in addition to common interventions. The outcomes, such as neck pain, cervical ROM, and functional limitations, were evaluated using a numeric pain rating scale (NPRS), standard universal goniometer, and neck disability index questionnaire at baseline and 4-week post-intervention. The paired and unpaired t-test was used to analyze the intervention effects on the outcomes within-group and between-group, keeping the significance level alpha set at p<0.05.

DETAILED DESCRIPTION:
The study hypothesised that adding the scapular functional training to the cervical isometric exercises will be equally effective than cervical isometric exercises alone on managing neck pain, cervical ROM, and functional limitations among participants with chronic mechanical neck pain. The present study is helpful for chronic mechanical neck pain patients and physiotherapist to better understand the effect of incorporation of the scapular functional training in the treatment of neck pain. Therefore, this protocol may be used as a treatment in chronic mechanical neck pain because it alleviates pain, neck disability, improving cervical range of motion in chronic mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female with aged range 22-35 years
* Neck pain of more than 3 months in duration
* Having neck pain without symptoms distal to shoulder
* Participant had not received any clinical treatment for their neck pain within 1-months, and
* Willingness to participate in the study.

Exclusion Criteria:

* Having a diagnosis of cervical spinal stenosis
* Patients with serious pathology (e.g., neoplasm, fractures and inflammatory diseases, unilateral and bilateral upper extremity radicular symptoms (cervical radiculopathy)
* Prior surgery of cervical spine
* Evidence of nerve root compression
* Pregnant women, and
* Showed poor cooperation in the study

Ages: 22 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
Neumeric pain rating scale (NPRS) | 4 weeks
  Neck pain was assessed by a nuemeric pain rating scale. It is an 11-points numeric scale marked with 0 to 10 between either end. Zero at one end and ten at the opposite end indicate no pain and unbearable/worst imaginable pain, respectively. The participants were asked to rate their current level of pain, as well as their worst and least amounts of pain in the past 24 hours.
Range of Motion (ROM) | 4 weeks
  Cervical range of motion was measured by a standard universal goniometer.
Functional limitations | 4 weeks
  The functional limitation due to mechanical neck pain was evaluated by a neck disability index questionnaire (NDI).

CONTACTS AND LOCATIONS:
Overall Officials: Amir Iqbal, MPT, Study Chair — King Saud University
Locations (1):
- Rehabilitation Research Chair, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Bharti N, Ahmed H, Hasan S, Iqbal A, Uddin S, Ahamed WM, Ahmad F, Mujtaba MA, Alghadir AH. Efficacy of Scapular Functional and Cervical Isometric Exercises in the Management of Chronic Mechanical Neck Pain: A Randomized Comparative Trial. Pain Res Manag. 2024 Dec 19;2024:5873384. doi: 10.1155/prm/5873384. eCollection 2024. PMID 39734604